CLINICAL TRIAL: NCT06792864
Title: Effectiveness of 3D Printed Polycaprolactone and Tricalcium Phosphate Bone Scaffold for Bone Regeneration in Cranioplasty: Randomized Clinical Trial
Brief Title: Effectiveness of 3D Bone Matrix in Cranioplasty
Acronym: OSTEOPRINTCR
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Austral de Chile (Other)
Responsible Party: Principal Investigator, Pedro C Aravena, PCAravena, Universidad Austral de Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORD541/2023
Record Dates: First submitted 2025-01-12; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Cranioplasty; Craniotomy; Craniotomy Clipping; Craniotomy Surgery; Craniocerebral Trauma; Craniocerebral Injuries
Keywords: Calcium Phosphates; Polyesters; Printing, Three-Dimensional; Skull / diagnostic imaging; Skull / surgery; Tissue Scaffolds
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- OsteoprintCR (Experimental): Hybrid technique of 3D printed bone scaffold based on polycaprolactone with beta-tricalcium phosphate
  Interventions: Device: OsteoprintCR
- SMAR SET GMV Endurance Gentamicin (Active Comparator): Patient submitted to cranioplasty with conventional technique using surgical cement based on polymethylmethylmethacrylate (PMMA) called "SMAR SET GMV Endurance Gentamicin".
  Interventions: Device: SMAR SET GMV Endurance Gentamicin

INTERVENTIONS:
Device: OsteoprintCR — Hybrid technique of 3D printed bone matrix based on polycaprolactone with tricalcium beta phosphate
  Arms: OsteoprintCR
Device: SMAR SET GMV Endurance Gentamicin — Patient undergoing cranioplasty with conventional technique using polymethylmethylmethacrylate-based surgical cement brand "SMAR SET GMV Endurance Gentamicin".
  Arms: SMAR SET GMV Endurance Gentamicin

SUMMARY:
The objective of this clinical trial is to evaluate the effectiveness of a 3D bone scaffold in relation to a scaffold formed by PCL + β-TCP (polycaprolactone and beta-tricalcium phosphate), compared to the use of PMMA (polymethyl methacrylate) acrylic cement for bone regeneration in patients undergoing cranioplasty in the city of Valdivia, Chile, between the years 2024-2025.

The main beneficiaries will be patients, users of the public or private health system, who require bone regeneration. The intermediate beneficiaries are the health team: doctors specialized in surgery and orthopedics, dedicated in their professional work to bone reconstruction and regeneration.

DETAILED DESCRIPTION:
The study will be a parallel-arm clinical trial (8 patients randomly divided into 2 groups), where the participants will be patients with cranial defects requiring cranioplasty at the Department of Neurosurgery of Base Hospital of Valdivia, Chile. Previously, data of each participant will be collected, such as sex, age, basic comorbidities and clinical diagnosis.

The outcome variables to be considered in this study are: The volume of bone reconstruction measure in axial computed tomography (CT) using the tool available in Mimics software delivering the value in cm3 , and the scaffold attachment to adjacent bone using the linear density scale in Hounsfield units (HU) where it will be considered from +3000 HU as dense bone formation and presence of GAP <1mm. The last variable will be the patients' perception of esthetics and quality of life, which will be measured using the "QOLIBRI" scale, where the items with the greatest difference in scores between the two groups will be highlighted; in addition, >80 total points will be considered as good quality of life.

Sample calculation: Considering the need to observe the maintenance of skull volume in functional and aesthetic aspects, according to the results of Park et al., the use of PCL/ß-TCP material observed a volume difference of 4.4 ± 2.5% at six months postoperatively versus the average initial volume, calculating the need for four study subjects per group (Effect size d= 1. 76; alpha error probability= 0.05; Power= 0.7; Allocation ratio N2/N1= 1. G*Power software U. Düsseldorf) An experimental group (PCL scaffold + β-TCP) and a control group (PMMA cement).

Surgical intervention PCL + β-TCP intervention protocol: Prior to surgery, the patient must answer a survey of concept of quality of life through the QOLIBRI guideline, followed by this the patient will undergo an initial CT scan where the necessary measurements of the bone defect will be performed to transfer this information to a graphic design software such as CAD 3D, the design and printing of the PCL + β-TCP segment will be performed in the Polymer Laboratory of the Universidad Austral de Chile, once obtained the digital files will be converted to a printable format (.gcode) compatible with fused deposition 3D equipment (FDM), using the Creality Ender-3 printer with PCL filament from Canada Filament Store with a diameter of 1.75 mm.

Subsequently, the prototype will be obtained where it will be verified that the graft has the required characteristics for each patient. Once this is approved, the sterilization protocol of the PCL+ß-TCP matrices will be carried out, which will be placed in a container with 70% ethanol and submerged for 15 minutes, after which time they will be placed on sterile absorbent paper to eliminate excesses. Finally, the scaffolds are exposed to UV light for 20 minutes. Finally, the matrices are packed. Then the surgery will be performed and a control CT scan will be taken 6 months after the intervention, together with the second QOLIBRI guideline.

PMMA surgical cement intervention protocol: The initial CT scan will be performed on each patient, then intraoperatively, the solid and liquid component of the PMAA cement will be mixed with enveloping movements until a homogeneous mass will be obtained that allows molding, With the surgical gloves moistened with physiological solution, the molding of the intraoperative PMMA platelet begins, taking the bone defect as a reference, looking for a thickness similar to the adjacent bone of the bone defect, previously, placing a latex patch (included with the PMMA prosthesis) protects the brain tissue. When the plate begins to increase its temperature during the exothermic polymerization process, it is removed from the surgical field and once the formed platelet is solid and cold, it is placed again in the bone defect, in order to adhere to the bone of the cranial calotte by means of a titanium fixation system. All patients are monitored in the intensive care unit for at least 24 hours in the immediate postoperative period, where a clinical and radiological (CT) follow-up will be performed to rule out ongoing clinical complications. Finally, a control CT scan will be taken 6 months after the intervention, together with the second QOLIBRI guideline.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 70 years of age, with acquired skull defect from neurological surgeries such as:

  * craniocerebral trauma,
  * refractory intracranial arterial hypertension,
  * congenital cranial defects such as hydrocephalus or other similar surgically resolvable defects,
* who are suitable for reconstruction using a PCL-TCP scaffold system;
* patients or their guardians are capable of giving valid informed consent.

Exclusion Criteria:

* Active infection at the time of study inclusion (in cases of chronic infection, active infections may manifest as a result of a failed trial of antibiotic withdrawal),
* immunodeficiency such as:

  * HIV,
  * systemic corticosteroid therapy,
  * chemotherapy,
  * synchronous hematologic malignancy,
  * other causes of secondary or primary immunodeficiency;
* patients with uncontrolled chronic diseases such ascardiovascular, respiratory or immunological diseases,
* psychiatric disorders not controlled with home pharmacotherapy,
* Women currently pregnant, breastfeeding or planning to become pregnant within 2 years of reconstruction surgery,
* patients with a life expectancy of less than 12 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Volume of bone reconstruction through computed tomography | 6 months
  Bone reconstruction volume: The CT scans (pre-surgery and 6 months post-surgery) will be compared using the Mimics software version 21.0 (Materialise NV, Leuven, Belgium) and the difference will be recorded in cm3.
Matrix bonding to the bone by computed tomography | 6 months
  The CT scans (pre-surgery and 6 months post-surgery) will be compared using the 3D Slicer software where specific areas of the tissue are selected, each pixel in the image has an associated density value that corresponds to a shade of gray which is known as the "Gray Scale" that discriminates the tissue densities in Hounsfield units (HU), a standardized scale based on the relative density of the tissues, comparing it with that of water (0 HU) and air (-1000 HU). Where it will be considered from +3000 HU as dense bone formation and presence of GAP <1mm.

SECONDARY OUTCOMES:
Perception of aesthetics and quality of life | 6 months
  Quality of life survey (QOLIBRI scale) which will be carried out in person in 2 instances of the study (before and after 6 months after surgery).
  The perception of quality of life will be measured with the QOLIBRI (Quality of Life after Brain Injury) guideline, which is validated and translated into Spanish, has 6 items and a score range from 0 to 100, where 100 is the highest quality of life. The items with the greatest difference in scores between the two groups will be highlighted; in addition, >80 total points will be considered as good quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Base de Valdivia, Valdivia, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hwang, K., Villavicencio, J.B. and Agdamag, A.M.P. (2021) 'Tissue Engineering and Regenerative Medicine Cranioplasty Using Polycaprolactone-Tricalcium Phosphate: Management and Treatment Outcomes', Neurosurgery Practice, 2(4), p. okab027. Available at: https://doi.org/10.1093/neuopn/okab027.
- [Result] Zubillaga Rodríguez, I., Sánchez Aniceto, G. and Montalvo Moreno, J.J. (2007) 'Reconstrucción craneal con biomateriales: Revisión histórica y estado actual', Revista Española de Cirugía Oral y Maxilofacial, 29(2), pp. 79-89.
- [Result] Park H, Choi JW, Jeong WS. Clinical Application of Three-Dimensional Printing of Polycaprolactone/Beta-Tricalcium Phosphate Implants for Cranial Reconstruction. J Craniofac Surg. 2022 Jul-Aug 01;33(5):1394-1399. doi: 10.1097/SCS.0000000000008595. Epub 2022 Mar 9. PMID 35261367
- [Result] Brachet A, Belzek A, Furtak D, Geworgjan Z, Tulej D, Kulczycka K, Karpinski R, Maciejewski M, Baj J. Application of 3D Printing in Bone Grafts. Cells. 2023 Mar 10;12(6):859. doi: 10.3390/cells12060859. PMID 36980200
- [Result] Gonzalez Matheus I, Hutmacher DW, Olson S, Redmond M, Sutherland A, Wagels M. A Medical-Grade Polycaprolactone and Tricalcium Phosphate Scaffold System With Corticoperiosteal Tissue Transfer for the Reconstruction of Acquired Calvarial Defects in Adults: Protocol for a Single-Arm Feasibility Trial. JMIR Res Protoc. 2022 Oct 13;11(10):e36111. doi: 10.2196/36111. PMID 36227628
- See also: A new method of cranioplasty — https://doi.org/10.3171/jns.1977.47.5.0790
- See also: Alloplastic Cranioplasty Reconstruction: A Systematic Review Comparing Outcomes With Titanium Mesh, Polymethyl Methacrylate, Polyether Ether Ketone, and Norian Implants in 3591 Adult Patients — https://journals.lww.com/annalsplasticsurgery/abstract/2019/05004/alloplastic_cranioplasty_reconstruction__a.4.aspx
- See also: Clinical Application of Three-Dimensional Printing of Polycaprolactone/Beta-Tricalcium Phosphate Implants for Cranial Reconstruction — https://journals.lww.com/jcraniofacialsurgery/fulltext/2022/07000/clinical_application_of_three_dimensional_printing.30.aspx
- See also: Craneoplastía con implante de polimetilmetacrilato (PMMA) para corregir secuela de trauma. Reporte de caso — https://revistas.unal.edu.co/index.php/actaodontocol/article/view/87341
- See also: Estudio de craneoplastía in situ empleando cemento de polimetilmetacrilato — https://www.ranc.com.ar/index.php/revista/article/view/592
- See also: Implantes personalizados de polimetilmetacrilato (PMMA) para aplicaciones en craneoplastia — https://repositorio.unal.edu.co/handle/unal/50398
- See also: Trauma craneoencefálico. Revisión de la literatura — https://www.revistachilenadeneurocirugia.com/index.php/revchilneurocirugia/article/view/82